CLINICAL TRIAL: NCT06846970
Title: The Effect of Adding Balneotherapy to the Physical Therapy Program on Neuropathic Pain, Disability, Daily Living Activities, and Sleep Quality in Patients with Chronic Lumbar Radiculopathy
Brief Title: Effects of Adding Balneotherapy to a Physical Therapy Program in Patients with Chronic Lumbar Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Betül Küçükdağ, Principal Investigator, MD, PhD, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTLLDH25
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Radiculopathy
Keywords: Chronic Lumbal Radiculopathy; balneotherapy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Physical Therapy and Balneotherapy (Experimental): Experimental: Physical Therapy and Balneotherapy Patients who received a conventional physical therapy and balneotherapy
  Interventions: Other: Experimental
- Active Comparator: Physical therapy only: Patients who received a conventional physical therapy (Active Comparator): Active Comparator: Physical therapy only: Patients who received a conventional physical therapy
  Interventions: Other: Active Comparator

INTERVENTIONS:
Other: Experimental — Patients will receive a conventional physical therapy program consisting of 20 sessions of exercise, hot pack, TENS, ultrasound and balneotherapy, five days a week and once a day for four weeks. Exercise, hot pack, TENS, ultrasound therapy, and balneotherapy will be performed under the supervision of a specialist physiotherapist.
  In both groups, patients will be evaluated by a physician at the beginning of the treatment, at the end of the 4-week treatment period, and at the 3rd month through clinical examination and assessment using the Visual Analog Scale (VAS), Oswestry Disability Index, Douleur Neuropathique 4 Questionnaire (DN4), Pain Quality Assessment Scale, LANSS (Leeds Assessment of Neuropathic Symptoms and Signs) Neuropathic Pain Scale, Short Form-36 (SF-36), and Pittsburgh Sleep Quality Index (PSQI).
  Arms: Experimental: Physical Therapy and Balneotherapy
Other: Active Comparator — Patients will receive a conventional physical therapy program consisting of 20 sessions of exercise, hot pack, tens and ultrosound therapy five days a week and once a day for four weeks. It was planned to perform exercise, hot pack, tens, ultrasound therapy accompanied by a specialist physiotherapist.
  In both groups, patients will be evaluated by a physician at the beginning of the treatment, at the end of the 4-week treatment period, and at the 3rd month through clinical examination and assessment using the Visual Analog Scale (VAS), Oswestry Disability Index, Douleur Neuropathique 4 Questionnaire (DN4), Pain Quality Assessment Scale, LANSS (Leeds Assessment of Neuropathic Symptoms and Signs) Neuropathic Pain Scale, Short Form-36 (SF-36), and Pittsburgh Sleep Quality Index (PSQI).
  Arms: Active Comparator: Physical therapy only: Patients who received a conventional physical therapy

SUMMARY:
The aim of this study is to investigate the effects of adding balneotherapy to the conventional physical therapy program on neuropathic pain, disability, daily living activities, and sleep quality in patients with chronic lumbar radiculopathy.

DETAILED DESCRIPTION:
Condition or Disease: Lumbar Radiculopathy, Neuropathic Pain, Disability, Daily Living Activities, Sleep Quality, Quality of Life Intervention/Treatment: Conventional Physical Therapy, Conventional Physical Therapy and Balneotherapy Phase: Not Applicable

Chronic lumbar radiculopathy is a clinical condition that occurs due to the compression of nerve roots in the lumbar region of the spinal cord, usually resulting from lumbar disc herniation, degenerative disc disease, spinal stenosis, or traumatic injuries. This condition leads to neuropathic pain and functional loss, significantly reducing patients' quality of life.

Neuropathic pain in chronic lumbar radiculopathy is characterized by symptoms such as burning, stinging, tingling, and electric shock-like sensations due to irritation or damage to the nerve roots. This type of pain may be difficult to manage with traditional analgesics and often requires a multidisciplinary treatment approach.

Balneotherapy is known to have analgesic, anti-inflammatory, and muscle-relaxant effects. In patients with chronic lumbar radiculopathy, balneotherapy has been shown to improve tissue oxygenation by increasing blood circulation, reduce muscle spasms, and regulate nerve functions. Additionally, it may enhance patients' functional capacity and participation in daily living activities.

Physical therapy is an effective method applied to reduce pain, increase muscle strength, and restore mobility in patients with chronic lumbar radiculopathy. Postural adjustments and manual therapy techniques can help alleviate nerve root compression and improve patients' quality of life. Modalities such as electrotherapy, ultrasound, and hot-cold applications may also be used to support treatment.

As a conclusion, a multidisciplinary treatment approach is necessary to control neuropathic pain and improve the quality of life and sleep quality of patients with chronic lumbar radiculopathy. The combination of balneotherapy and physical therapy may be effective in alleviating symptoms and enhancing functional capacity. Further clinical research is needed to more comprehensively determine the effectiveness of these treatment methods.

In this study, patients aged 18-75 years who have been diagnosed with chronic lumbar radiculopathy based on history, physical examination, clinical findings, lumbar MRI, and EMG results will be included. One group will receive a physical therapy program, while the other group will receive both a physical therapy program and balneotherapy.

Both groups will be assessed at baseline, after four weeks of treatment, and at the third month through physician evaluations and examinations. The study will employ scales such as the Visual Analog Scale (VAS), Oswestry Disability Index, Douleur Neuropathique 4 Questionnaire (DN4), Pain Quality Assessment Scale, LANSS (Leeds Assessment of Neuropathic Symptoms and Signs) Neuropathic Pain Scale, Short Form-36 (SF-36), and Pittsburgh Sleep Quality Index (PSQI) to investigate whether adding balneotherapy to a physical therapy program affects neuropathic pain, disability, daily living activities, and sleep quality in patients with chronic lumbar radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years who have been diagnosed with chronic lumbar radiculopathy based on medical history, physical examination, clinical findings, lumbar MRI, and EMG results, and who present to the outpatient clinic for physical therapy without any contraindications for treatment, will be included in the study after obtaining their informed consent.

Exclusion Criteria:

* Patients with thermoregulation disorders or sensory deficits
* Patients with lesions that impair skin integrity
* Patients with decompensated heart failure
* Patients with advanced heart, liver, or kidney failure
* Patients with advanced, uncontrolled peripheral venous insufficiency
* Patients with a history of epilepsy or seizures
* Patients with pregnancy, malignancy, or a recent surgical operation
* Patients in the acute exacerbation phase of rheumatic diseases
* Patients with severe anemia
* Patients with tuberculosis
* Patients with febrile infectious diseases
* Patients with diseases associated with bleeding disorders
* Patients who have undergone regular balneotherapy in the past three months
* Patients with polyneuropathy or peripheral nerve damage
* Patients with muscle weakness detected during examination
* Patients with prostheses
* Patients with a history of lumbar surgery Exclusion Criteria for Balneotherapy
* Patients with thermoregulation disorders or sensory deficits
* Patients with lesions that impair skin integrity
* Patients with decompensated heart failure
* Patients with advanced heart, liver, or kidney failure
* Patients with advanced, uncontrolled peripheral venous insufficiency
* Patients with a history of epilepsy or seizures
* Patients with pregnancy, malignancy, or a recent surgical operation
* Patients in the acute exacerbation phase of rheumatic diseases
* Patients with severe anemia
* Patients with tuberculosis
* Patients with febrile infectious diseases
* Patients with diseases associated with bleeding disorders
* Patients who have undergone regular balneotherapy in the past three months
* Patients with polyneuropathy or peripheral nerve damage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Visuel Analog Scale (VAS) | Time Frame: Baseline, after 4 weeks and 3 months
  The musculoskeletal pain intensity of the patients is assessed using the Visual Analog Scale (VAS). The meanings of the numbers placed on a 10 cm line ranging from 0 to 10 are explained to the patients. A score of 0 indicates no pain, 10 represents the most severe pain ever experienced, and 5 is explained as moderate pain. Based on this explanation, patients are asked to rate their pain levels by considering the past week.
Change in Oswestry Disability Index (ODI) | Time Frame: Baseline, after 4 weeks and 3 months
  Oswestry Disability Index is a crucial tool used to assess the severity of low back pain and functional impairment. It is widely utilized in clinical practice, research, and treatment planning. The questionnaire evaluates ten different categories of activities that affect participants' daily lives. These categories include walking, sitting, standing, rising, sleeping, personal care, and the ability to perform work-related tasks. Participants are asked to rate each activity on a specific scale. The results are calculated as a percentage
Change in Douleur Neuropathique 4 Questionnaire (DN4) | Time Frame: Baseline, after 4 weeks and 3 months
  DN4 is a short-form questionnaire designed to detect and diagnose neuropathic pain symptoms. The questionnaire consists of 10 questions that assess the symptoms experienced by the patient, specifically targeting characteristics associated with neuropathic pain. A score ranging from 0 to 10 is assigned based on the responses.
Change in LANSS Neuropathic Pain Assessment Scale | Time Frame: Baseline, after 4 weeks and 3 months
  To determine the presence of neuropathic pain, all patients will be assessed using the Self-Administered Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) Scale. The S-LANSS scale is designed to differentiate neuropathic pain from nociceptive pain. Unlike the standard LANSS scale, the S-LANSS does not require a physician's physical examination, making it easier to administer.
  The S-LANSS scale consists of seven questions, which are self-reported by the patient. The first five questions assess pain-related symptoms, while the last two questions involve self-applied clinical examination. Responses are yes/no, with different point values assigned to each question. The total score is 24, and a score of 12 or higher suggests the presence of neuropathic pain. The Turkish version of the S-LANSS scale has been validated for reliability and accuracy.

SECONDARY OUTCOMES:
Change in Pain Quality Assessment Scale (PQAS) | Time Frame: Baseline, after 4 weeks and 3 months
  The Pain Quality Assessment Scale is commonly used to evaluate the characteristic features of pain. These features include pain description (e.g., sharp, burning, stabbing), pain distribution (localized, widespread), accompanying symptoms (e.g., swelling, redness), and pain duration (acute, chronic). A scoring system ranging from 0 to 10 is applied for each question. This scale is widely used in clinical settings, pain research, and pain management planning.
Change in Short Form-36 (SF-36) | Time Frame: Baseline, after 4 weeks and 3 mo
  The Short Form-36 (SF-36) Health Survey is a generic self-administered quality of life assessment tool consisting of 36 items. It has been validated for reliability and validity in patients with musculoskeletal disorders. The SF-36 measures eight dimensions of health-related quality of life:
  * Physical Functioning (10 items)
  * Social Functioning (2 items)
  * Role Limitations due to Physical Problems (3 items)
  * Mental Health (5 items)
  * Energy/Vitality (4 items)
  * Pain (2 items)
  * General Health Perceptions (5 items) The SF-36 assesses both positive and negative aspects of health status, considering the past four weeks. In six of the eight dimensions, patients are asked to rate their status on a three- or six-point scale. The scores for each domain are coded and converted into a scale ranging from 0 (worst health status) to 100 (best health status).
Change in Pittsburgh Sleep Quality Index (PSQI) | Time Frame: Baseline, after 4 weeks and 3 months
  The Pittsburgh Sleep Quality Index is a self-reported questionnaire designed to evaluate sleep quality over the past four weeks. It consists of 24 items that assess various aspects of sleep. The PSQI includes seven components, each scored on a scale of 0 to 3. The total PSQI score ranges from 0 to 21, with scores above 5 indicating poor sleep quality. The Turkish version of the PSQI has been validated for reliability and accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Bestas Bestas, Principal Investigator, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (2):
- Turkey (Türkiye) (2):
  - Afyonkarahisar HSU, Afyonkarahisar, Afyonkarahisar, Central
  - Afyonkarahisar HSU, Afyonkarahisar, Central

REFERENCES:
- [Background] Dilekci E, Ozkuk K, Kaki B. The short-term effects of balneotherapy on pain, disability and fatigue in patients with chronic low back pain treated with physical therapy: A randomized controlled trial. Complement Ther Med. 2020 Nov;54:102550. doi: 10.1016/j.ctim.2020.102550. Epub 2020 Sep 4. PMID 33183668
- [Background] Onat SS, Tasoglu O, Guneri FD, Ozisler Z, Safer VB, Ozgirgin N. The effectiveness of balneotherapy in chronic low back pain. Clin Rheumatol. 2014;33(10):1509-15. doi: 10.1007/s10067-014-2545-y. Epub 2014 Mar 6. PMID 24599676
- [Background] Dogan M, Sahin O, Elden H, Hayta E, Kaptanoglu E. Additional therapeutic effect of balneotherapy in low back pain. South Med J. 2011 Aug;104(8):574-8. doi: 10.1097/SMJ.0b013e318224644f. PMID 21886066